CLINICAL TRIAL: NCT02842606
Title: Effects of the Consumption of Fiber-enriched Pasta on Glucose and Lipid Metabolism and Satiety
Brief Title: Metabolic Response to the Acute Consumption of Fiber-enriched Pasta
Acronym: PROPASTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, rivellese angela, Full professor, Federico II University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 166/14
Record Dates: First submitted 2016-07-15; First posted 2016-07-25 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2016-07

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fiber-enriched pasta (Experimental): The participants consume whole wheat pasta with added fiber (fiber 12 g fiber/100 g).
  Interventions: Other: Test meal
- Control pasta (Active Comparator): The participants consume pasta made from durum wheat semolina (fiber 2.7g/100g).
  Interventions: Other: Test meal

INTERVENTIONS:
Other: Test meal — The two test meals are designed to have the same energy and macronutrient composition. They differ only in the carbohydrate source: fiber-enriched pasta or control pasta. Blood samples are taken at fasting and every 30 minutes over 4 hours. Fasting and postprandial intestinal fermentation is evaluated by breath test.
  Other Names: Acute test meal

SUMMARY:
Cardio-metabolic diseases are a leading cause of mortality worldwide. Over the years, therefore, there have been considerable efforts to identify strategies for prevention and management of risk factors. The diet, with its pleiotropic effects, is one of the most effective approaches to reduce the cardio-metabolic risk. In this context, the dietary fibers have been extensively studied and the available evidence supports the beneficial effects of its consumption. However, worldwide the average fiber consumption is still less than the recommended daily dose. For this reason, the availability of functional foods, such as additional sources of fiber in the diet, may facilitate the attainment of fiber recommended.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18-29 kg / m2
* Good Health status

Exclusion Criteria:

* Diabetes
* Cardiovascular events (IMA or stroke) severe heart disease
* Kidney or liver failure
* Anemia and any other chronic disease

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-03; Primary Completion 2015-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Glucose and lipid response | 4 hours
  Evaluated by enzymatic colorimetric methods

SECONDARY OUTCOMES:
Insulin response | 4 hours
  Evaluated by ELISA
Hormone response (GLP-1, GIP, PYY and Ghrelin) | 4 hours
  Evaluated by ELISA
Energy intake in the subsequent meal. | 4 hours
  Evaluated by food record

IPD SHARING:
Plan to Share IPD: No